CLINICAL TRIAL: NCT03622216
Title: A Dose Escalation Study to Assess the Efficacy and Safety of Bradanicline in Subjects With Refractory Chronic Cough
Brief Title: A Dose Escalation Study of Bradanicline in Refractory Chronic Cough
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Attenua, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ATA101-PN-001
Record Dates: First submitted 2018-08-02; First posted 2018-08-09 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Chronic Cough
MeSH Terms: conditions — Chronic Cough

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bradanicline QD (Experimental): Randomized crossover design of 3 different doses of bradanicline (film-coated tablets) to be administered orally QD
  Interventions: Drug: Bradanicline; Drug: Placebo
- Placebo (Placebo Comparator): Randomized crossover design of matching placebo tablets to be administered orally QD
  Interventions: Drug: Bradanicline; Drug: Placebo

INTERVENTIONS:
Drug: Bradanicline — Three different doses over the course of the study
Drug: Placebo — Matching placebo for Bradanicline

SUMMARY:
This is a randomized, double-blind, placebo-controlled, crossover, dose escalation study of bradanicline in subjects with chronic cough

DETAILED DESCRIPTION:
This study will have two 21-day treatment periods separated by a 14-day washout period. There will be a 14-day follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Chest radiograph or computed tomography (CT) scan of the thorax within the last 1 year not demonstrating any abnormality considered to be significantly contributing to the refractory chronic cough
* Diagnosis of refractory chronic cough or unexplained cough for at least one year
* Women of child-bearing potential who use 2 forms of acceptable birth control method
* Male subjects and their partners of child-bearing potential who use 2 methods of acceptable birth control
* Has provided written informed consent

Exclusion Criteria:

* Current smoker (cigarettes or e-cigarettes) or has given up smoking within the past 12 months
* Currently taking an ACE-inhibitor or requiring treatment with an ACE-inhibitor during the study or within 12 weeks prior to the Baseline Visit
* Has an upper or lower respiratory tract infection or recent significant change in pulmonary status within 4 weeks of the Baseline Visit
* Has a history of cystic fibrosis
* Has a history of malignancy within 5 years prior to the Baseline Visit
* Has active hepatitis infection
* Has a history of human immunodeficiency virus (HIV) infection
* Has a positive test for any drug of abuse
* Has a history of hypersensitivity to bradanicline or any of its components

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
Awake coughs per hour at Days 7, 14, 21, 43, 50, 57 | Change from Baseline at Days 7, 14, 21, 43, 50, 57
  Assessment of awake coughs per hour (average hourly cough frequency while the participant is awake based on sound recordings), to be evaluated using a digital recording device

SECONDARY OUTCOMES:
24-hour coughs per hour at Days 7, 14, 21, 43, 50, 57 | Change from Baseline at Days 7, 14, 21, 43, 50, 57
  Assessment of 24-hour coughs per hour (average hourly cough frequency based on 24-hour sound recordings), to be evaluated using a digital recording device
Percentage of participants who have at least one adverse event (AE) during the treatment periods, washout, and follow-up | up to 57 days
  Assessment of participants who have at least one AE during treatment period 1 (21 days), during washout (14 days), during treatment period 2 (21 days), and follow-up (14 days)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Attenua, Inc.
Locations (17):
- United States (17):
  - BioSolutions Clinical Research Center, La Mesa, California
  - Allergy & Asthma Associates of Southern California, Mission Viejo, California
  - Asthma and Allergy Associates, Colorado Springs, Colorado
  - Storms Clinical Research Institute, Colorado Springs, Colorado
  - Colorado Allergy and Asthma Center, Denver, Colorado
  - Center for Cough, Largo, Florida
  - Florida Pulmonary Research Institute, Winter Park, Florida
  - Clinical Research Institute, Plymouth, Minnesota
  - Mayo Clinic, Pulmonary Clinic Research Unit, Rochester, Minnesota
  - Atlantic Research Center, LLC, Ocean Township, New Jersey
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - National Allergy and Asthma Research, North Charleston, South Carolina
  - AARA Research Center, Dallas, Texas
  - Pharmaceutical Research and Consulting, Inc., Dallas, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Bellingham Asthma Allergy and Immunology Clinic, Bellingham, Washington
  - Allery Asthma & Sinus Center, Greenfield, Wisconsin